CLINICAL TRIAL: NCT05774041
Title: Visualization of the STN and GPi for DBS Surgery in Patients With Parkinson's Disease
Brief Title: Visualization of the STN and GPi for DBS
Acronym: VISION
Status: Terminated | Type: Observational
Why Stopped: Study terminated by Sponsor
Sponsor: Surgical Information Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOC-0039
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Deep Brain Stimulation; Parkinson Disease
Keywords: Subthalamic nucleus; Globus pallidus; DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SIS Group: Standard of care DBS surgery + use of (FDA-cleared) SIS System for preoperative target planning
  Interventions: Device: SIS System
- Control Group: Standard of care DBS surgery and preoperative target planning

INTERVENTIONS:
Device: SIS System — FDA-cleared software that enhances standard clinical images for the visualization of structures in the basal ganglia area of the brain which are commonly targeted for DBS lead placement.
  Groups: SIS Group

SUMMARY:
The purpose of the study is to determine if using SIS System for DBS planning results in less distance between the planned target location and the actual implanted lead location than DBS planning without SIS System.

DETAILED DESCRIPTION:
This is a prospective, controlled, open-label, multicenter post-market trial to compare standard of care DBS surgery to standard of care plus visualization with the SIS System. The purpose of the study is to determine if using SIS System for DBS planning results in less distance between the planned target location and the actual implanted lead location than DBS planning without SIS System.

Parkinson's Disease subjects indicated for DBS will undergo standard DBS surgery with preoperative planning for targeting of STN or GPi as indicated. Subjects will be followed through six months after initial DBS programming to collect clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with Idiopathic Parkinson's Disease and is indicated for de novo DBS surgery with bilateral DBS leads implanted in the STN or GPi.
* Subject is 18 years or older.
* Subject must be able and willing to provide informed consent and comply with study follow-up schedule and procedures.

Exclusion Criteria:

* Subject is not a DBS surgical candidate due to untreated, clinically significant depression, current suicidal ideation, or dementia or any neuropsychological condition or finding that would contraindicate DBS surgery.
* Subject had prior intracranial surgery or other implanted neurostimulators or drug delivery pumps.
* Subject's life expectancy is less than one year.
* Subject is Hoehn and Yahr stage 4-5 in the medication OFF condition.
* Subject is pregnant or interested in becoming pregnant during the duration of the study.
* Subject is currently enrolled in another clinical study utilizing investigational medications, devices, or treatment that would conflict with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic Parkinson's Disease indicated for de novo bilateral DBS surgery implant in the STN or GPi will be considered for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Measure Euclidean distance (mm) between the planned target coordinate and actual implanted coordinate | 1 day
  Compare the mean distance between the DBS planned target location to the actual implanted lead location for the SIS Group and Control Group

OTHER OUTCOMES:
Proportion of patients(%) with procedure-related adverse events, average duration of DBS surgery (hours:minutes), and percentage of cases in which intra-operative testing was performed | 1 month
  Compare surgical characteristics, such as rate of procedure-related adverse events, mean surgical time, and use of intra-operative testing for SIS and Control groups
Compare width of the therapeutic window (the electrical current at which a sustained side effect occurs minus the electrical current at which a meaningful therapeutic benefit was observed) | 6 months
  Compare DBS programming settings, such as therapeutic window of SIS and Control groups
Change in average levodopa equivalent daily dosage (mg) | 6 months
  Compare change in mean levodopa equivalent daily dose for SIS and Control groups
Change in mean score of the Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III | 6 months
  Compare changes in mean MDS-UPDRS Part III motor improvement for SIS and Control groups. MDS-UPDRS Part III is a validated questionnaire to assess the severity of motor symptoms in patients with Parkinson's disease. The motor examination consists of 33 scored movements. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score is obtained from the sum of the corresponding item scores.
Rate (%) of stimulation-related side effects | 6 months
  Compare the rate of stimulation related side effects in SIS and Control groups
Compare percentage of motor benefit from MDS-UPDRS Part III to implanted lead location | 6 months
  Measure hemi-body motor improvement and compare percentage of improvement to the implanted DBS lead location

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Hartford Hospital, Hartford, Connecticut
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Penn State University, Hershey, Pennsylvania
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No